CLINICAL TRIAL: NCT06469411
Title: The Effect MSCs Derived From the Placenta and Their Secretome for the Treatment of GvHD: A Randomized Clinical Trial
Brief Title: Effect of PMSCs and Their Secretome for the Treatment of GvHD
Acronym: GvHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tabriz University of Medical Sciences (Other)
Collaborators: SCARM Institute, Tabriz, Iran (Other Government)
Responsible Party: Principal Investigator, Abolfazl Barzegari, Principal Investigator, SCARM Institute, Tabriz, Iran
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRCT20201108049311N7; 71647 (Other Grant/Funding Number: Tabriz University of Medical Sciences)
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: GVHD
Keywords: Bone marrow; Mesenchymal stem cell; Secretome; Severe Graft-versus-host disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Secretome

STUDY DESIGN:
Intervention Model Description: In this clinical trial study, 60 patients with GvHD, who were referred to Shahid Qazi Hospital in Tabriz, were randomly divided into 2 groups of 30 people, and the intervention and control groups received secretome and distilled water by injection, respectively. The method of blinding was tripleblinded and all the names and personal information of the patients was coded at the time of data collection and remain completely confidential.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was a triple-blinded study. In this way, the doctor introduced the patients to receive secretome/distilled water and was not aware of the grouping. Participating volunteers did not know about receiving secretome, distilled water, or other drugs. Secretome and distilled water were placed in similar and coded vials. In addition, the placebo (distilled water) was identical in appearance (shape and color), taste, and smell with secretome. In addition, due to the coding of patients and the lack of clarity in the grouping of patients, the data analyzer were be also blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Recipient of 6 doses secretome (set of substances released from the cell to its surroundings) of mesenchymal stem cells retrieved from the placenta (containing 400 microgram protein/ milliliter) (It was produced through the cell culture from the placenta in the laboratory) 4 cc dissolved in albumin 20% every week for 6 weeks
  Interventions: Biological: Secretome (set of substances released from the cell to its surroundings) of mesenchymal stem cells retrieved from the placenta (containing 400 microgram protein/ milliliter)
- Control group (Placebo Comparator): Recipient of 6 doses of 4 cc distilled water dissolved in albumin 20% every week for 6 weeks
  Interventions: Other: 4 cc distilled water dissolved in albumin 20%

INTERVENTIONS:
Biological: Secretome (set of substances released from the cell to its surroundings) of mesenchymal stem cells retrieved from the placenta (containing 400 microgram protein/ milliliter) — Patients in the intervention arm received 6 doses of secretome of mesenchymal stem cells retrieved from the placenta (containing 400 microgram protein/ milliliter) 4 cc dissolved in albumin 20% every week for 6 weeks
  Arms: Intervention group
Other: 4 cc distilled water dissolved in albumin 20% — Patients in the control arm received 6 doses of 4 cc distilled water dissolved in albumin 20% every week for 6 weeks
  Arms: Control group

SUMMARY:
In this clinical trial study, 60 patients with GvHD referred to Shahid Qazi Hospital in Tabriz, were randomly divided into 2 intervention and control groups (n= 30 in each) that received secretome and distilled water by injection, respectively. The method of blinding was triple-blinded and all the names and personal information of the patients were coded at the time of data collection and remained completely confidential.

DETAILED DESCRIPTION:
This study is a safety, feasibility, and efficacy trial that was conducted on eligible GvHD patients with the diagnosis of expert doctors after obtaining permission from the respected ethics committee and registering the trial at the Iranian Trial Registration Center. During the phone call, while stating the title and objectives of the study, the entry and exclusion criteria were checked. If they are eligible, they were asked to attend the Ghazi Hospital if they wish to participate in the study. In the face-to-face meeting, the objectives of the research were fully explained and the study criteria were re-examined. The written informed consent was obtained and questionnaires fulfilled three times which include personal-social characteristics, medical characteristics, appetite questionnaire, 24-hour food record (Food record), and family members. At the beginning of the study, 50 cc of blood was used to collect serum and to culture and condition mesenchymal stem cells. 200 men with GvHD were randomly assigned using random block method using blocks of 4 and 6 and RAS (Random Allocation Software) and allocation ratio 1:1 to two groups receiving intravenous secretome with The first protocol (30 people) and receiving the mesenchymal stem cells secretome of the second protocol (30 people) were allocated and they received the skin spray for 1 year. Participants in the first protocol group at the beginning of the study, day 3, end of the week, the end of the second week, and the end of the month 5 times and in the second protocol group at the beginning of the study, skin spray were done. The secretome of both groups was the same.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute GvHD with fever and requiring hospitalization

Exclusion Criteria:

* Patients with sepsis

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Liver involvement | At the beginning of the study and 6 weeks after the intervention
  Measurement of Bilirubin level
Intestine condition | At the beginning of the study and 6 weeks after the intervention
  Diarrhea volume measurement
Skin rash | At the beginning of the study and 6 weeks after the intervention
  Determination of BSA percentage

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Ghasemi Moghadam, MD, Principal Investigator — Stem Cell and Regenerative Medicine Institute, Tabriz University of Medical Sciences, Tabriz, Iran; Sepideh Zununi Vahed, PhD, Study Director — Kidney Research Center, Tabriz University of Medical Sciences, Tabriz, Iran; Babak Nejati, MD, Study Director — Hematology and Oncology Research Center, Tabriz University of Medical Sciences, Tabriz, Iran; Graciela Pavon-Djavid, PhD, Study Chair — Université Sorbonne Paris Nord, INSERM U1148, Laboratory for Vascular Translational Science, Cardiovascular Bioengineering, 99 Av. Jean-Baptiste Clément 93430 Villetaneuse, France
Locations (1):
- Abolfazl Barzegari, Tabriz, East Azerbaijan Province, Iran